CLINICAL TRIAL: NCT05592249
Title: The Effect of Different Dual Task Practices on Activities of Daily Living in Stroke Individuals
Brief Title: The Effect of Dual Tasks on ADL in Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Ayse Zengin Alpozgen, Asst. Prof. (PhD), Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 10.2022
Record Dates: First submitted 2022-10-20; First posted 2022-10-24 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Stroke; Dual Task; Activity of Daily Living
Keywords: Activity; Hemiplegia; Cognitive
MeSH Terms: conditions — Stroke; Motor Activity; Hemiplegia

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Motor - Cognitive (Experimental): Motor - Cognitive group will receive motor and cognitive dual task intervention.
  Interventions: Other: Dual Task MC
- Motor - Motor (Experimental): Motor - Motor group will receive motor and motor dual task intervention.
  Interventions: Other: Dual Task MM

INTERVENTIONS:
Other: Dual Task MC — Dual Task MC group will receive 60 minutes motor - cognitive dual task intervention 5 day per week for 6 weeks in clinic.
  Arms: Motor - Cognitive
Other: Dual Task MM — Dual Task MM group will receive 60 minutes motor - motor dual task intervention 5 day per week for 6 weeks in clinic.
  Arms: Motor - Motor

SUMMARY:
The aim of this study is to investigate the effectiveness of different dual-task practices on activities of daily living in stroke patients. The sample size was calculated as 18 people for each group and 36 people in total, with a 20% drop out. MC (Motor - Cognitive) group will receive 60 minutes motor - cognitive dual task intervention 5 day per week for 6 weeks in clinic. MM (Motor - Motor) group will receive 60 minutes motor - motor dual task intervention 5 day per week for 6 weeks in clinic. As the primary outcomes in the study; Modified Barthel Index will be used to evaluate basic activities of daily living, Nottingham Extended Activities of Daily Living Index designed specifically for stroke to evaluate instrumental activities of daily living, and Stroke Impact Scale 3.0 to evaluate participation in activities of daily living. As secondary outcomes; 10 Meter Walk Test will be used for functional mobility assessment, Timed Up and Go Test and Berg Balance Scale will be used for balance assessment, Motor Activity Log-28 will be used to assess upper extremity functions, and Montreal Cognitive Assessment Test will be used for cognitive status assessment.

DETAILED DESCRIPTION:
Postural control is lost due to decrease in unilateral muscle strength and joint range of motion, and increase in muscle tone in stroke individuals, and accordingly, deterioration in balance and coordination between the two sides of the body is observed. Spasticity, abnormal movement patterns, and loss of motor control are observed in patients, and ambulation limitations occur in patients. In addition, approximately two-thirds of stroke patients have impairments in cognitive skills, which are necessary for the realization of motor skills. Depending on the executive dysfunction, problems also arise in the planning, sequencing, and coordination of actions. Stroke patients have difficulty in doing many activities that they encounter in their daily lives, such as walking and climbing stairs, and as a result, their quality of life and participation in daily life activities are negatively affected. For this reason, approaches aimed at regulating not only muscle tone and strength, but also approaches to ensure participation in daily life activities and increase functionality should be preferred in the rehabilitation process of stroke patients.

Considering the traditional approaches applied in stroke rehabilitation, it is seen that balance and gait training are frequently given to patients. However, in daily life, it may be necessary to use cognitive skills as well as motor activities simultaneously or to perform two motor skills at the same time. Patients have difficulty in performing two tasks at the same time, such as carrying a bag while climbing stairs, calculating while walking, and reading a newspaper while on an exercise bike. In order to increase the participation of stroke patients in daily life, the dual-task approach should be included in the treatment strategies.

Dual task applications are the ability to perform two tasks at the same time, which have different goals and can be evaluated separately, and is a motor learning-based approach. One of the tasks may be a motor task and the other may be a cognitive task, or both may be a motor task. Studies have concluded that dual-task training has positive effects on gait parameters, balance, and cognition, and it has been reported that it is a current approach that can be used in the treatment of stroke patients. However, there is no study comparing the participation of dual tasks, such as one cognitive and one motor task or two motor tasks, in activities of daily living in stroke patients.

When activities of daily living are examined, most of the motor activities are accompanied by actions that include cognitive processes such as attention, memory, problem solving, and concentration. For this reason, in this study, it is assumed that different dual-task approaches to be applied in the rehabilitation of stroke patients will give different results in the participation of individuals in daily life activities and that the application of motor and cognitive tasks together will be more effective than the application of two motor tasks together. In the light of all these, the aim of this study is to investigate the effectiveness of different dual-task practices on activities of daily living in stroke patients.

The hypothesis of this study is;

H0: In the dual task approach applied to individuals with stroke, the application of motor and cognitive tasks together is not more effective in daily living activities compared to the two motor tasks.

H1: In the dual task approach applied to individuals with stroke, the application of motor and cognitive tasks together is more effective in daily living activities compared to the two motor tasks.

ELIGIBILITY:
Inclusion Criteria:

* To be diagnosed with stroke by a specialist physician
* Modified Rankin Score ≤ 3 with moderate or mild disability
* To score 21 and above on the Montreal Cognitive Assessment Test
* Be over 18 years old
* Volunteering to participate in the study

Exclusion Criteria:

* Presence of additional neurological disease
* Having orthopedic problems that may prevent walking
* Presence of apraxia
* The patient has a hearing loss that cannot understand the commands given
* To have a score below 30 on the Beck Depression Scale

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2022-12-26 (Actual); Primary Completion 2023-12-20 (Actual); Study Completion 2024-02-20 (Actual)

PRIMARY OUTCOMES:
Modified Barthel Index | 6 weeks
  The Modified Barthel Index (MBI) is a scale created to evaluate functional independence. The scale evaluates the functional independence level of the person in 10 activities, including transfer, ambulation, stairs, feeding, dressing, personal care, bathroom, toilet use, and urine and stool continence. Each question is answered in 5 different levels. Level 1 means "The individual is inadequate to do the activity." while Level 5 means "Completely independent.". The score that the patient can get is between 0-100. The higher the score, the higher the person's level of functional independence.
Nottingham Extended Activities of Daily Living Index | 6 weeks
  The Nottingham Extended Activities of Daily Living Index is a scale designed specifically for stroke and evaluated by self-report. This scale, which aims to measure the quality of daily life of individuals in instrumental activities based on performance, consists of 4 subgroups as movement, kitchen, housework and leisure activities and a total of 22 items. Each question evaluates the difficulty of the activity on a 4-point Likert scale. 0 points means "I can't do it at all." 3 points means "I do it easily by myself.". The maximum score that can be obtained from the scale is 66. An increase in the score indicates independence in the instrumental activities of daily living.
Stroke Impact Scale 3.0 | 6 weeks
  The Stroke Impact Scale (SIS) 3.0 aims to evaluate the quality of life of patients after stroke, consists of 8 subsections and a total of 59 questions. It evaluates muscle strength, hand functions, activities of daily living, mobility, communication skills, mood, memory and participation of patients after stroke. Each question is scored by evaluating on a 5-point Likert-type scale. 1 point means not being able to perform the function asked at all, while 5 points means not having any difficulties. In addition to 8 sub-sections, there is a visual analog scale that is scored between 0-100 at the end of the scale and the perception of recovery after stroke is evaluated. A score of 0 on this scale is "No improvement at all." A score of 100 means "Complete recovery". The maximum score that can be obtained is 395, and the minimum score is 59. An increase in the total score in SIS indicates the independence of the patient in activities of daily living while a decrease indicates dependence.

SECONDARY OUTCOMES:
10 Meter Walk Test | 6 weeks
  The 10 Meter Walk Test (10 MWT) is a test that evaluates a person's walking performance. For the application, a total distance of 14 meters is determined with the start and end points of which the first and last 2 meters are marked. The patients are asked to walk the determined distance at their normal walking speed, and as soon as the 2 meter line is reached, the measurement is started with the stopwatch, and the stopwatch is stopped at the 12 meter line. The time is recorded in seconds. To minimize effects such as habituation and fatigue, the test is repeated twice and the average second is recorded. In stroke patients, if the gait speed is below 0.4 m/s, it is interpreted as indoor ambulation, between 0.4-0.8 m/s as limited community ambulation, and above 0.8 m/s as full community ambulation.
Timed Up and Go Test | 6 weeks
  The Timed Up and Go Test (TUG) is a general physical performance test used to evaluate a person's balance and locomotor performance. The assessment ends with the person getting up from the chair, walking 3 meters, turning around, and returning to sit on the chair again. The person is told to walk at a normal walking pace. The time is recorded in seconds. Completing the test in less than 10 seconds is interpreted as being completely independent, completing the test between 10-20 seconds is considered independent for main transfers, and completing the test over 30 seconds is interpreted as needing help in most activities.
Berg Balance Scale | 6 weeks
  Berg Balance Scale (BBS) is a 14-item scale that measures the ability of individuals to maintain their balance during functional activities. Each task in the scale is scored between 0-4. 0 point means "Cannot perform independently." 4 point means "Completes the activity independently.". The maximum score that can be obtained from the scale is 56. A score of 0-20 indicates balance disorder and high fall risk, 21-40 points indicates the presence of an acceptable balance and moderate fall risk, 41-56 points indicates the presence of good balance and low fall risk.
Motor Activity Log - 28 | 6 weeks
  The Motor Activity Log - 28 (MAL - 28) consists of two scales questioning how often the patient uses the upper extremity on the affected side during various activities and, if so, with what quality. The person answers the questions on the scale by scoring between 0 and 5. 0 point means "I don't use my affected arm at all." 5 point means "I use my affected arm in the same way as before the stroke.". If the patient has difficulty in scoring, he can also use half points such as 2.5, 3.5. If the patient chooses 0 points during scoring, the reason is questioned and one of the 5 reasons for not using is noted. The maximum score that can be obtained from the scale is 280. The higher the score, the higher the frequency and quality of use of the arm.
Montreal Cognitive Assessment Test | 6 weeks
  MOCA is an assessment scale used to evaluate cognitive impairment. It includes items evaluating visuospatial skills, executive functions, naming, memory, attention, language, abstract thinking, delayed recall, and orientation. The maximum score that can be obtained from the scale is 30, and the minimum score is 0. Scores of 21 and above are considered normal. A decrease in the score indicates cognitive impairment in the patient.

CONTACTS AND LOCATIONS:
Overall Officials: Ayşe Zengin Alpözgen, Asst. Prof., Principal Investigator — Istanbul University - Cerrahpasa
Locations (1):
- Istanbul University - Cerrahpasa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No